CLINICAL TRIAL: NCT07112105
Title: Repetitive Transcranial Magnetic Stimulation Treatment of Stimulant Use Disorder
Acronym: VA-StARTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRD4-003-24W; 1-I01-RD-000693-01-A2 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stimulant Use Disorder
Keywords: Magnetic resonance imaging; Transcranial magnetic stimulation; Intermittent theta burst stimulation; Dopamine; Reward processing
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups to receive active or sham rTMS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which participants, staff administering treatment, investigators, and outcome assessors are all masked to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Experimental): Receive active rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS (Sham Comparator): Receive sham rTMS
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — rTMS is a non-invasive procedure in which administering a transient magnetic field induces electrical currents in specific, targeted brain regions. The intervention (active and sham) will be administered in 30 sessions across 2 weeks. The brain region targeted is the dorsolateral prefrontal cortex.
  Arms: Active rTMS
Device: Sham rTMS — Subjects randomized to sham rTMS will undergo the same procedures on the same equipment as subjects assigned to active rTMS, but no active magnetic stimulation will be delivered.
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to establish a new treatment (repetitive transcranial stimulation (rTMS)) for Veterans with stimulant use disorder (SUD). Despite the large public health burden imposed by SUD, there is currently no FDA-approved or widely recognized effective somatic treatment. This placebo controlled study will test the effectiveness of rTMS in the treatment of SUD, and explore biomarkers that may guide patient selection for rTMS treatment and predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for DSM Disorders (SCID) confirmed diagnosis of SUD, severe
* Last use of stimulants >2 and <8 weeks
* Stable medication regimen (no change in dose or agents between 2 weeks prior to the start of and throughout the treatment phase of the study)
* Stable medical health

Exclusion Criteria:

* Pregnant or lactating female
* History of prior adverse reaction to TMS
* On medications thought to significantly lower seizure threshold, e.g. clozapine, chlorpromazine, clomipramine, and bupropion > 400mg/day
* Seizure disorder or conditions known to substantially increase risk for seizures
* Implants or medical devices incompatible with TMS
* Acute or unstable chronic medical illness that would affect participation or compliance in the study, e.g. unstable angina
* Unstable psychiatric symptoms that precludes consistent participation in the study, e.g. active current suicidal intent or plan; severe psychosis
* Other substance use disorder not in remission
* Chronic or recurring Axis I psychotic disorders
* For subjects participating in fMRI scans, presence of ferromagnetic material in their body or taking DAergic medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Relapsed | 3 months after last rTMS treatment
  Rate of stimulant use relapse compared between active vs. sham rTMS groups

SECONDARY OUTCOMES:
Reward circuit function and signaling | Within 1 week before rTMS treatment and within 1 week after rTMS treatment
  Before and after treatment, participants will undergo functional magnetic resonance imaging (fMRI) imaging while completing the Monetary Incentive Delay Task, a validated probe of reward processing circuit function and dysfunction. Signaling in the substantia nigra will be measured in an individual-subject, "native space" region of interest approach as a marker of dopaminergic reward processing function, as well as in voxel-wise, whole-brain exploratory analyses. Changes in reward function and signaling will be compared between active vs. sham rTMS groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jong H. Yoon, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No